CLINICAL TRIAL: NCT05029102
Title: TAS-102 Combined With Anlotinib in Patients With Metastatic Gastric Cancer Refractory to Standard Treatments (THALIA): a Prospective Single-arm Phase II Study
Brief Title: TAS-102 and Anlotinib in ≥3 Lines mGC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weijia Fang, MD, Director of Medical Oncology, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THALIA
Record Dates: First submitted 2021-08-29; First posted 2021-08-31 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — trifluridine tipiracil drug combination; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAS-102 and Anlotinib (Experimental): TAS-102: 35 mg/m2，per oral，twice daily, days 1-5 and 8-12 of each 28-day cycle Anlotinib: 10mg，per oral，once daily，days 1-14 of each 21-day cycle
  Interventions: Drug: TAS 102; Drug: Anlotinib

INTERVENTIONS:
Drug: TAS 102 — 35 mg/m2，per oral，twice daily, days 1-5 and 8-12 of each 28-day cycle
Drug: Anlotinib — 10mg，per oral，once daily，days 1-14 of each 21-day cycle

SUMMARY:
To determine the efficacy and safety of TAS-102 and Anlotinib in patients with metastatic gastric cancer who had been treated with ≥ 2 lines of prior standard chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, ≤75 years
* Histologically confirmed gastric cancer with distant metastasis
* ECOG 0-1
* Progression on ≥ 2 lines of prior standard chemotherapy
* Patients can swallow pills normally
* Expected overall survival ≥6 months
* Blood routine: no blood transfusion or blood products usage within 14 days, G-CSF or other hematopoietic stimulator was not used. WBC counts > 3000/µl，Absolute neutrophil count (ANC) ≥ 1500 cells/µl，Platelet count ≥ 100,000/µl，Hemoglobin ≥ 9.0 g/dL.
* AST, ALT and alkaline phosphatase ≤ 2.5 times the upper limit of normal (ULN)，Serum bilirubin ≤ 1.5 x ULN，creatinine<ULN
* Prothrombin time (PT), international standard ratio (INR) ≤1.5 × ULN
* Women of childbearing age must be willing to use adequate contraceptives during the study period of drug treatment;
* Informed consent has been signed.

Exclusion Criteria:

* Active bleeding within 3 months; Occurrence of arterial/venous thrombosis within 6 months; Hereditary or acquired bleeding (e.g., clotting dysfunction) or thrombotic tendencies; Full dose oral or injectable anticoagulants or thrombolytic drugs for therapeutic purposes are currently being used or have been used recently (10 days prior to the commencement of study treatment); Surgery (except for biopsy) was performed within 4 weeks prior to the study or the surgical incision was not fully healed; Aspirin (> 325 mg/ day) or dipyridamole, ticlopidine, clopidogrel, and silotazole are currently being used or have recently been used (10 days prior to the study).
* Certain or suspected brain metastases.
* Patients who have received prior therapy of any study drug;
* Serious uncontrolled systemic diseases, such as severe active infections;
* A person is known to be infected with the immunodeficiency virus (HIV) or known to be HIV-positive;
* Patients have suffered from other malignancies in the past 5 years except cervical carcinoma in situ or basal cell carcinoma of the skin
* Untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers (HBV DNA >500 IU/mL) or active HCV carriers with HCV RNA can be detected. Remarks: Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B patients (HBV DNA < 500 IU/mL) may be enrolled
* Anti-infective therapy was not discontinued 14 days before the study;
* A prior history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonia, and symptomatic interstitial lung disease or the presence of active pneumonia on a chest CT scan within 4 weeks prior to the study.
* Patients have a history of intestinal obstruction within six months. Patients with incomplete obstruction syndrome of ileus at the time of initial diagnosis may be enrolled in the study if they have received definitive (surgical) treatment to resolve the symptoms, as assessed by the investigator.
* Patients have high blood pressure that cannot be well controlled by antihypertensive medication (systolic ≥140 mmHg or diastolic ≥90 mmHg)
* Urine routine indicated urinary protein ≥++ and confirmed 24-hour urinary protein >1.0g;
* Known to be allergic to any study drug;
* Patients have participated in other drug clinical studies within 4 weeks before enrollment;
* Lactating women
* According to the judgment of the researcher, the patient may have other factors that may affect the results of the study or cause the study to be terminated, such as alcohol abuse, drug abuse, other serious diseases (including mental diseases) requiring combined treatment. Patients have severe laboratory abnormalities, which will affect the safety of the patient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 4 months
  The time elapsed between treatment initiation and tumor progression

SECONDARY OUTCOMES:
Overall Response Rate | 2 months
  the proportion of patients in a trial whose tumor is destroyed or significantly reduced by a drug. ORR is generally defined as the sum of complete responses (CRs) - patients with no detectable evidence of a tumor over a specified time period - and partial responses (PRs) - patients with a decrease in tumor size over a specified time period.
Overall Survival | 9 months
  Refers to the time of death from enrollment to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- First affiliated hospital, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ying T, Xia R, Zhang Y, Dai J, Wang Y, Xie X. Cost-effectiveness analysis of trifluridine/tipiracil in the treatment of heavily pretreated metastatic gastric cancer from the perspective of Chinese healthcare system. BMJ Open. 2024 Nov 7;14(11):e080846. doi: 10.1136/bmjopen-2023-080846. PMID 39510786